CLINICAL TRIAL: NCT04695054
Title: Combined Use of Buzzy and EMLA Cream for Vascular Access in Children. A Randomized Controlled Trial
Brief Title: Buzzy Plus EMLA Cream for Vascular Access in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 12/2019
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Vascular Access
Keywords: Children; Buzzy device; EMLA cream; Peripheral vascular access

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buzzy and EMLA Cream (Experimental): In the experimental group children will receive the application of EMLA cream 60 minutes before the needle procedure and the use of Buzzy device during the procedure.
  Interventions: Device: Buzzy device plus EMLA cream
- EMLA Cream (Active Comparator): In the control group children will receive the application of EMLA cream 60 minutes before the needle procedure
  Interventions: Drug: Only EMLA cream

INTERVENTIONS:
Device: Buzzy device plus EMLA cream — EMLA cream will be applied 60 minutes before the needle procedure; the Buzzy device will be used during the procedure
  Arms: Buzzy and EMLA Cream
Drug: Only EMLA cream — EMLA cream will be applied 60 minutes before the needle procedure
  Arms: EMLA Cream

SUMMARY:
Venepuncture and peripheral intravenous cannulation are commonly performed in children and may cause substantial pain and distress. The aim of this study is to evaluate the efficacy of the combination of EMLA cream and Buzzy device in pain and distress relief during venipuncture or peripheral vascular access in hospitalized children.

The study is an open randomized controlled study. Eligible children will be randomized to receive the application of EMLA cream 60 minutes before the needle procedure or the application of EMLA 60 minutes before the procedure and the use of Buzzy device during procedure.

The primary study outcome will be the mean distress score experienced by children at the moment of the procedure, evaluated with the CEMS scale. Secondary outcomes will be the mean distress score recorded by operators; the self-reported mean pain score; the mean pain score reported by parents and operators.

ELIGIBILITY:
Inclusion Criteria:

* children between 4 and 12yrs of age needing venipuncture or peripheral vascular access
* children who have applied EMLA cream at least 60 minutes before the procedure

Exclusion Criteria:

* children with cognitive impairment
* children with skin lesion that does not allow the application of Buzzy device
* children diseases that cause hypersensibility to cold (i.e. Raynaud syndrome, sickle cell disease)
* children who have taken any analgesics in the 8 hours before enrollment

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Mean distress evaluated by parents | Intraprocedural
  Distress score will be recorded by parents through the use of the Children's Emotional Manifestation Scale (CEMS scale). The CEMS scale is an observational scale validated for recording procedural distress in children. It takes into consideration the following characteristics: facial expression, vocalization, activity, interaction, cooperation, with a score ranging from a minimum of 5 (no distress) to a maximum of 25 (serious distress)

SECONDARY OUTCOMES:
Mean distress evaluated by operators | intraprocedural
  Distress score will be recorded through the use of the Children's Emotional Manifestation Scale (CEMS scale). The CEMS scale is an observational scale validated for recording procedural distress in children. It takes into consideration the following characteristics: facial expression, vocalization, activity, interaction, cooperation, with a score ranging from a minimum of 5 (no distress) to a maximum of 25 (serious distress)
Mean pain score evaluated by children | Immediately after the procedure
  Pain scores will be reported through the Faces Pain Scale Revised (FPS-R scale). The FPS-R algometric scale is appropriate for the detection of pain in children aged 4 to 12 years, as it includes both a series of smiley faces with an expression that changes according to increasing pain, and a numerical scale, for a pain scale ranging from zero (no pain) to 10 (severe pain).
Mean pain score evaluated by parents | Immediately after the procedure
  Pain scores will be reported through the Faces Pain Scale Revised (FPS-R scale). It includes both a series of smiley faces with an expression that changes according to increasing pain, and a numerical scale, for a pain scale ranging from zero (no pain) to 10 (severe pain).
Mean pain score evaluated by operators | Immediately after the procedure
  Pain scores will be reported through the Faces Pain Scale Revised (FPS-R scale). It includes both a series of smiley faces with an expression that changes according to increasing pain, and a numerical scale, for a pain scale ranging from zero (no pain) to 10 (severe pain).
Success at first attempt | Intraprocedural
  Percentage of success of the procedure on the first attempt in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Strajn, Nurse, Principal Investigator — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (1):
- IRCCS materno infantile Burlo Garofolo, Trieste, TS, Italy